CLINICAL TRIAL: NCT02223208
Title: Romidepsin in Combination With CHOEP as First Line Treatment Before Hematopoietic Stem Cell Transplantation in Young Patients With Nodal Peripheral T-cell Lymphomas: a Phase I-II Study
Brief Title: Ro Plus CHOEP as First Line Treatment Before HSCT in Young Patients With Nodal Peripheral T-cell Lymphomas
Acronym: FIL_PTCL13
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_PTCL13
Record Dates: First submitted 2014-07-21; First posted 2014-08-22 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Peripheral T-cell Lymphomas (PTCL); PTCL-NOS; Angioimmunoblastic T-cell Lymphoma (AITL); ALK- Anaplastic Large Cell Lymphoma (ALCL); Nodal Peripheral T-Cell Lymphoma of T Follicular Helper Cell Origin
Keywords: PTCL; PTCL-NOS; AITL; ALCL
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Immunoblastic Lymphadenopathy | interventions — Clinical Trials, Phase I as Topic; romidepsin; Cyclophosphamide; Doxorubicin; Vincristine; Etoposide; Prednisone; Clinical Trials, Phase II as Topic

ARMS (1):
- Ro-CHOEP-21 (Experimental): During the Phase I It will administered Romidepsin (dose escalation) and the combination of CHOEP-21. During the Phase II It will administered Romidepsin (dose according to phase I) and the combination of CHOEP-21.
  Interventions: Drug: Ro-CHOEP-21 (PHASE I); Drug: Ro-CHOEP-21 (PHASE II)

INTERVENTIONS:
Drug: Ro-CHOEP-21 (PHASE I) — Romidepsin (dose escalation) Starting dose: 12mg/ms iv day +1 and +8
  Dose modification according to toxicity:
  * 14mg/ms day +1 and +8
  * 10mg/ms day +1 and +8
  * 8mg/ms day +1 and +8
  CHOEP-21
  * Doxorubicin 50 mg/ms iv day +1 or +2,
  * Vincristin 1.4 mg/ms (maximum 2.0 mg total dose) iv day+1 or +2
  * Cyclophosphamide 750 mg/ms iv day +1 or +2
  * Etoposide 100mg/ms iv from day +1 to +3 or from day +2 to +4
  * Prednisone100 mg orally from days +1 to +5 or from days +2 to +6
  PR or CR:Ro-CHOEP-21 for 3 additional cycles followed by stem cell mobilization and transplantation phase (CR --> AUTO-SCT, PR --> ALLO-SCT)
  Other Names: Romidepsin; Cyclophosphamide; Doxorubicin; Vincristin; Etoposide; Prednisone
Drug: Ro-CHOEP-21 (PHASE II) — Ro-CHOEP-21 x 3 cycles
  * Romidepsin dose according to phase I iv day +1 and +8
  * Doxorubicin 50 mg/ms iv day +1 or +2,
  * Vincristin 1.4 mg/ms (maximum 2.0 mg total dose) iv day+1 or +2,
  * Cyclophosphamide 750 mg/ms iv day +1 or +2
  * Etoposide 100mg/ms iv from day +1 to +3 or from day +2 to +4
  * Prednisone100 mg orally from days +1 to +5 or from days +2 to +6
  PR or CR: Ro-CHOEP-21 for 3 additional cycles followed by stem cell mobilization and transplantation phase (CR --> AUTO-SCT, PR --> ALLO-SCT)
  Other Names: Romidepsin; Cyclophosphamide; Doxorubicin; Vincristin; Etoposide; Prednisone

SUMMARY:
This is a multicenter study that includes two phases:

1. A phase I study to define the maximum tolerated dose (MTD) of Romidepsin in addition to CHOEP-21 and to test the safety and feasibility of CHOEP-21 in combination with dose escalation of Romidepsin (8, 10, 12, 14 mg). The dose level defined as MTD of Romidepsin will be used for the subsequent phase II study.
2. A phase II study to evaluate the efficacy (response rate, progression free survival and overall survival) and safety of Ro-CHOEP-21 incorporated into a treatment strategy including SCT.

DETAILED DESCRIPTION:
PHASE I A1) Induction phase Ro-CHOEP-21 x 3 cycles

* Romidepsin (dose escalation) starting dose: 12mg/ms iv day +1 and +8. Dose modification according to toxicity (14mg/ms day +1 and +8; 10mg/ms day +1 and +8; 8mg/ms day +1 and +8);
* CHOEP-21 (Doxorubicin 50 mg/ms iv day +1; Vincristin 1.4 mg/ms (maximum 2.0 mg total dose) iv day+1; Cyclophosphamide 750 mg/ms iv day +1; Etoposide 100mg/ms iv from day +1 to +3; Prednisone100 mg orally from days +1 to +5).

According to the response achieved after the first 3 Ro-CHOEP-21 cycles:

* PR or CR: Ro-CHOEP-21 for 3 additional cycles followed by phase A2
* SD or PD: Treatment failures, proceed to salvage according to each institutional policy.

A2) Stem cell mobilization and transplantation phase Response evaluation and one DHAP course followed by peripheral stem cell harvesting.

According to response achieved after 6 Ro-CHOEP-21 cycles:

CR: BEAM or FEAM or CEAM followed by auto-SCT PR

* Allogeneic SCT with HLA-identical (A, B, C, DR, DQ loci) or one antigen mismatched (class I) sibling donors. Donor selection is based on molecular high-resolution typing (4 digits) of the HLA gene loci class I (HLA-A, B, and C) and class II (DRB1, DQB1). In case, no class I and class II completely identical urelated donor (10 out of 10 gene loci) can be identified, the degree of histocompatibility between patient and donor must fulfill with the minimal degree of matching established by the Italian Bone Marrow Donor Registry: HLA-A and HLA-B antigen histocompatibility and HLA-DRB1 allelic histocompatibility.
* when a suitable donor is not available: BEAM or FEAM or CEAM followed by Auto-SCT.
* Haploidentical transplantation is allowed in selected cases < PR: Treatment failures, proceed to salvage according to each institutional policy.

PHASE II A1) Induction phase Ro-CHOEP-21 x 3 cycles

* Romidepsin dose according to phase I iv day +1 and +8
* Doxorubicin 50 mg/ms iv day +1,
* Vincristin 1.4 mg/ms (maximum 2.0 mg total dose) iv day+1,
* Cyclophosphamide 750 mg/ms iv day +1,
* Etoposide 100mg/ms iv from day +1 to +3
* Prednisone100 mg orally from days +1 to +5

According to the response achieved after the first 3 Ro-CHOEP-21 cycles:

* PR or CR: Ro-CHOEP-21 for 3 additional cycles followed by phase A2
* SD or PD: Treatment failures, proceed to salvage according to each institutional policy.

A2) Stem cell mobilization and transplantation phase Response evaluation and one DHAP course followed by peripheral stem cell harvesting.

According to response achieved after 6 Ro-CHOEP-21 cycles:

CR: BEAM or FEAM or CEAM followed by auto-SCT PR

* Allogeneic SCT with HLA-identical (A, B, C, DR, DQ loci) or one antigen mismatched (class I) sibling donors. Donor selection is based on molecular high-resolution typing (4 digits) of the HLA gene loci class I (HLA-A, B, and C) and class II (DRB1, DQB1). In case, no class I and class II completely identical urelated donor (10 out of 10 gene loci) can be identified, the degree of histocompatibility between patient and donor must fulfill with the minimal degree of matching established by the Italian Bone Marrow Donor Registry: HLA-A and HLA-B antigen histocompatibility and HLA-DRB1 allelic histocompatibility.
* when a suitable donor is not available: BEAM or FEAM or CEAM followed by Auto-SCT.
* Haploidentical transplantation is allowed in selected cases < PR: Treatment failures, proceed to salvage according to each institutional policy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 e ≤ 65 years
2. Peripheral T-cell lymphomas at diagnosis including: PTCL-NOS, AITL including other nodal TFH, ALK-ALCL
3. Stage II-IV
4. Written informed consent
5. No prior treatment for lymphoma
6. No Central Nervous System (CNS) disease (meningeal and/or brain involvement by lymphoma)
7. HIV negativity
8. Absence of active hepatitis C virus (HCV) infection
9. HBV negativity or patients with HBcAb +, HBsAg -, HBs Ab+/- with HBV-DNA negativity (in these patients Lamivudine prophylaxis is mandatory)
10. Levels of serum bilirubin, alkaline phosphatase and transaminases < 2 the upper normal limit, if not disease related
11. No psychiatric illness that precludes understanding concepts of the trial or signing informed consent
12. Ejection fraction > 50% and myocardial stroke in the last year nor QT prolongation (QTc interval < 480 msec using the Fridericia formula)
13. Clearance of creatinine > 60 ml/min if not disease related
14. Spirometry Diffusion Capacity (DLCO) > 50%
15. Absence of active, uncontrolled infection
16. For males and females of child-bearing potential, agreement upon the use of effective contraceptive methods prior to study entry, for the duration of study participation and in the following 90 days after discontinuation of study treatment
17. Availability of histological material for central review and pathobiological studies.

Exclusion Criteria:

1. Age <18 e > 65 years
2. Hystology other than: PTCL-NOS, AITL, ALK-ALCL
3. Stage I
4. Prior treatment for lymphoma
5. Positive serologic markers for human immunodeficiency virus (HIV)
6. Active hepatitis B virus (HBV) infection
7. Active hepatitis C virus (HCV) infection
8. Levels of serum bilirubin, alkaline phosphatase and transaminases > 2 the upper normal limit, if not disease related
9. Ejection fraction < 50% and no myocardial stroke in the last year or QT prolongation (QTc interval > 480 msec using the Fridericia formula)
10. Clearance of creatinine < 60 ml/min if not disease related
11. Spirometry Diffusion Capacity (DLCO) < 50%
12. Pregnancy or lactation
13. Patient not agreeing to take adequate contraceptive measures during the study
14. Psychiatric disease that precludes understanding concepts of the trial or signing informed consent
15. Any active, uncontrolled infection
16. Prior history of malignancies other than PTCLs in the last five years (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) of Ro-CHOEP-21 (Phase I endpoint) | 3 months
  Incidence of dose-limiting toxicity (DLT) of Ro-CHOEP-21, considering as maximum dose the one causing induction of any grade ≥ 3 non hematologic toxicity or a delay >15 days of planned cycle date observed during the first two cycles according to the definitions of NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 (2009)
Progression Free Survival (PFS) of Ro-CHOEP-21 (Phase II endpoint) | 18 months
  PFS on intention to treatment (ITT) evaluated at 18 months. PFS will be defined as the time between the date of enrolment and the date of disease progression, relapse or death from any cause.

SECONDARY OUTCOMES:
Proportion of patients reaching SCT (Phase I endpoint) | 6 months
  Proportion of patients reaching SCT
ORR = Overall response rate (Phase I endpoint) | 6 months
  Overall response rate (ORR, defined according to the Cheson 2007 response criteria) of the combination of Ro-CHOEP-21.
Overall Response Rate (ORR) and Complete Response (CR)(Phase II endpoint) | 6 months
  ORR and CR (defined according to the Cheson 2007 response criteria), after induction treatment and after SCT.
Event free survival (EFS) (Phase II endpoint) | 18 months
  Event free survival (EFS) defined as the time between the date of enrollment and the date of discontinuation of treatment for any reason
Overall survival (OS) (Phase II endpoint) | 24 months
  Overall survival (OS) defined as the time between the date of enrolment and the date of death from any cause in the ITT population enrolled in the study
Progression Free Survival (PFS) and Overall Survival (OS) (Phase II endpoint) | 3 months
  PFS and OS in patients not responding to the first 3 courses of Ro-CHOEP-21
Toxicities (Phase II endpoint) | 18 months
  Evaluation during the interim analyses of any grade III or higher toxicities, recorded and classified according to the definitions of NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 (2009)
Higher toxicities (Phase II endpoint) | 18 months
  Evaluation during all the pretransplant phase of any grade III or higher toxicities, recorded and classified according to the definitions of NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 (2009)
Treatment-related mortality (TRM) (Phase II Endpoint) | 24 months
  Treatment-related mortality defined as any death that was not attributable to the lymphoma.
Graft-versus-host disease (GVHD) (Phase II endpoint) | 24 months
  Incidence of acute and chronic GVHD in allografted patients

OTHER OUTCOMES:
Evaluation of response biomarkers (eg TET2 mutations) | 8 years
  Evaluation of response biomarkers (eg TET2 mutations)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Corradini, Prof, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano
Locations (27):
- Italy (27):
  - Ospedale SS. Antonio e Biagio e Cesare Arrigo, Alessandria, AL
  - Policlinico S. Orsola Malpighi, Bologna, BO
  - Spedali Civili, Brescia, BS
  - Ospedale Businco, Cagliari, CA
  - Azienda Ospedaliera S.Croce e Carle, Cuneo, CN
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.) - Sede di Meldola, Meldola, FC
  - IRCCS AOU San Martino - Clinica Ematologica, Genova, GE
  - IRCCS AOU San Martino - UO Ematologia 1, Genova, GE
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, MI
  - Fondazione IRCCS "Istituto Nazionale dei Tumori", Milan, MI
  - Azienda Ospedaliera Ospedale Niguarda Ca' Granda, Milan, MI
  - AO Ospedali Riuniti Villa Sofia - Cervello (Presidio Cervello), Palermo, PA
  - IRCCS Centro di Riferimento Oncologico (CRO), Aviano, PN
  - AOU di Parma, Parma, PR
  - Fondazione IRCCS - Policlinico San Matteo, Pavia, PV
  - IRCCS Arcispedale "Santa Maria Nuova", Reggio Emilia, RE
  - Ospedale degli Infermi, Rimini, RN
  - AO Città della Salute e della Scienza - Ematologia 1U, Torino, TO
  - AO Città della Salute e della Scienza - SC Ematologia, Torino, TO
  - AOU "Santa Maria della Misericordia", Udine, UD
  - Ospedale Borgo Roma, Verona, VR
  - Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale, Napoli
  - Ospedale Maggiore della Carità - SCDU Ematologia, Novara
  - A.O. di Perugia - Santa Maria della Misericordia, Perugia
  - Ospedale G. Da Saliceto - AUSL di Piacenza, Piacenza
  - UO Ematologia Ospedale S.Maria delle Croci, Ravenna